CLINICAL TRIAL: NCT04878068
Title: POC Study to Evaluate the Performance of the Therma COVID-19 Rapid Antigen Test for Detection of SARS-CoV-2 Virus in Human Saliva
Brief Title: Study to Evaluate the Performance of the Therma COVID-19 Rapid Antigen Test for Detection of SARS-CoV-2
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cannabis Research Associates (Other)
Responsible Party: Sponsor
Other Study IDs: TB20
Record Dates: First submitted 2021-04-27; First posted 2021-05-07 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-04

CONDITIONS: Covid19
Keywords: Saliva Antigen; Rapid Saliva Test
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Rapid Antigen Saliva Test: Participants who have had a COVID-19 PCR test will self-administer the saliva test. The research team will conduct the processing of the test for the results of positive, negative or inconclusive
  Interventions: Device: Theram COVID-19 Rapid Antigen Test

INTERVENTIONS:
Device: Theram COVID-19 Rapid Antigen Test — The Therma COVID-19 Rapid Antigen Test is an in vitro rapid, lateral flow immunoassay intended for the qualitative detection of SARS-CoV-2 nucleocapsid protein antigens in human saliva specimens. This test is intended for near-patient use at the point-of-care or lay person, self-use in a non-laboratory or home setting using saliva samples from individuals with or without symptoms of COVID-19.

SUMMARY:
The Therma COVID-19 Rapid Antigen Test is an in vitro rapid, lateral flow immunoassay intended for the qualitative detection of SARS-CoV-2 nucleocapsid protein antigens in human saliva specimens. This test is intended for near-patient use at the point-of-care or lay person, self-use in a non-laboratory or home setting using saliva samples from individuals with or without symptoms of COVID-19.

The Therma COVID-19 Rapid Antigen Test will be compared to a Health Canada approved RT-PCR COVID-19 test. Nasopharyngeal (for RT-PCR) samples will be collected at a COVID-19 Testing centre and saliva (for the rapid antigen test) samples will be collected and compared.

The prospective, observational, feasibility study will test 300 participants to establish the performance characteristics of the test on saliva specimens.

ELIGIBILITY:
Inclusion Criteria:

1. Participant is willing to sign verbal informed consent form
2. Age 12 or older and parents or legal guardians must consent for children as required by law.
3. Participant is attending COVID-19 testing centre for a nasopharyngeal swab sample
4. Participant is willing to provide a self-collected saliva sample

Exclusion Criteria:

1. Participant has previously tested positive for COVID-19 within the past 90 days

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Potential participants attending a COVID-19 testing centre for a PCR test will be approached to determine eligibility and obtain consent after they have had their PCR test completed. Three hundred participants will be recruited into the study.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2021-05-15 (Estimated); Primary Completion 2021-06-30 (Estimated); Study Completion 2021-06-30 (Estimated)

PRIMARY OUTCOMES:
Establish Performance of Therma COVID-19 Rapid Antigen Test | 1 day
  To establish the performance characteristics of the Therma COVID-19 Rapid Antigen Test in a near-patient, point-of-care (POC) setting with lay users (no laboratory experience) testing a participant that has self-collected the saliva specimen. Clinical accuracy of the rapid antigen test compared to RT-PCR test results. Accuracy refers to the (PPA, positive percent agreement (sensitivity) and (NPA, negative percent agreement (specificity) between the results of the tests. The expected performance of the test for symptomatic participants shall be >90% PPA and >98% NPA.

SECONDARY OUTCOMES:
Participant Feedback | 1 day
  Evaluate participant feedback on the usability of the Therma COVID-19 Rapid Antigen Test and saliva collection device using the Participant Study Questionnaire Form (Ease of use 5-point scale from 5=Easy to 1=Hard)
User Feedback | 1 day
  Evaluate user feedback on the usability of the Therma COVID-19 Rapid Antigen Test and saliva collection device using the Therma Feasibility Study User Feedback Questionnaire (ease of use 5-point scale from Not at all to Very easy)

CONTACTS AND LOCATIONS:
Overall Officials: Ira Price, MD, Principal Investigator — McMaster University